CLINICAL TRIAL: NCT06103357
Title: Identification of Innovative Circulating and Cellular Biomarkers in Subjects With Acute and Chronic Coronary Syndrome (PLAQUE Study)
Brief Title: Identification of Biomarkers in Subjects With Coronary Syndrome (PLAQUE Study)
Acronym: PLAQUE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: INRCA_009_2023
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-10

CONDITIONS: Coronary Syndrome
Keywords: Acute Coronary Syndrome; Chronic Coronary Syndrome; microRNAs; soluble ST2; interleukin-6
MeSH Terms: conditions — Angina, Unstable; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects with clinical indication for coronary angioplasty: Twenty subjects with acute or chronic coronary syndrome that will be underwent to angioplasty procedure according to standard clinical practice.
  Interventions: Other: blood sample collection

INTERVENTIONS:
Other: blood sample collection — Before and after angioplasty, blood samples upstream and downstream of the coronary lesion will be taken, arterial sampling at the aortic root level will be performed, and peripheral venous blood will be collected.

SUMMARY:
The study will to test the levels of innovative biomarkers, such as miRNAs, in the blood of subjects underwent to angioplasty procedure according to standard clinical practice.

DETAILED DESCRIPTION:
Twenty patients with acute coronary syndrome from non-ST-segment elevation myocardial infarction or with chronic coronary syndrome with clinical indication and favorable anatomy for coronary angioplasty will be enrolled. The angioplasty procedure will be performed according to standard clinical practice. Before and after angioplasty, blood samples will be taken upstream and downstream of the coronary lesion, arterial sampling will be performed at the level of the aortic root, and peripheral venous blood will be collected. MicroRNA expression will be analyzed in serum by next-generation sequencing (miRNome). Quantitative analysis of pro- and anti-inflammatory molecules such as IL-6 and the soluble form of IL-33 receptor (sST2) will be performed on various blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for the PCI procedure according to the latest ESC (European Society of Cardiology) Guidelines
* Coronary stenosis treated with angioplasty must be located in the proximal segments of the three main vessels: IVA, CX and CD
* The vessels must have a diameter of their mid-distal section ≥ 3 mm
* Patients with NSTEMI ACS and clinical indication with favorable anatomy for coronary angioplasty, also called percutaneous coronary intervention (PCI), (for the ACS group)
* Patients with clinically incipient SCC with stable angina (or significant anginal equivalents) and clinical indication with favorable anatomy for PCI (for the SCC group)

Exclusion Criteria:

* Contraindications to anticoagulant/antiplatelet therapy
* Extensive calcifications and/or tortuosity of the major epicardial segments
* Evidence of thrombotic occupation
* Patients with hemodynamic instability
* Patients with EF (ejection fraction) < 35%
* Patients with severe chronic renal failure (e-GFR < 30 mL/min)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by Acute Coronary Syndrome (ACS) and Chronic Coronary Syndrome (CCS) with clinical indications for coronary angiography, demonstrating the presence of significant coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
miRNome analysis | baseline
  The Next Generation Sequencing (NGS) techniques will be used to identify miRNome picture as potential biomarkers for acute and chronic coronary syndrome.

SECONDARY OUTCOMES:
Identification of biomarkers of inflammation | baseline
  Interleukin-6 and soluble ST2 levels will be assessed in plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Antonicelli, MD, Study Director — IRCCS INRCA
Locations (1):
- IRCCS INRCA Hospital, Ancona, Italy

REFERENCES:
- [Derived] Protic O, Bonfigli AR, Olivieri F, Lamedica AM, Gabrielli G, Antonicelli R. miRNome profile in blood samples upstream and downstream of the coronary lesion and arterial aortic root before and after angioplasty in subjects with chronic and acute coronary syndrome: A pilot observational study protocol (Plaque study). PLoS One. 2025 Jun 13;20(6):e0324467. doi: 10.1371/journal.pone.0324467. eCollection 2025. PMID 40512691